CLINICAL TRIAL: NCT03787810
Title: Left Ventricular Dysfunction in Critically Ill Patients
Acronym: LEVEDYCIP
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Jonatan Oras, Consultant, adjunct senior lecturer, Sahlgrenska University Hospital
Other Study IDs: LEVEDYCIP
Record Dates: First submitted 2018-12-23; First posted 2018-12-26 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2019-09

CONDITIONS: Left Ventricular Dysfunction; Critically Ill; Acute Coronary Syndrome; Cardiomyopathies; Takotsubo Cardiomyopathy
MeSH Terms: conditions — Ventricular Dysfunction, Left; Critical Illness; Acute Coronary Syndrome; Cardiomyopathies; Takotsubo Cardiomyopathy | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography — Echocardiography for assessment of left ventricular dysfunction

SUMMARY:
Left ventricular dysfunction is common in the critically ill. The aim of this study is to assess the incidence and prognosis of left ventricular dysfunction in critically ill patients.

DETAILED DESCRIPTION:
Left ventricular dysfunction is common in the critically ill. A number of conditions can cause left ventricular dysfunction including myocardial infarction, septic cardiomyopathy, post resuscitation syndrome, takotsubo syndrome etc. A number of studies have assessed cardiac dysfunction in specific conditions (e.g. sepsis, cardiac arrest) but only a few studies have assessed cardiac dysfunction in a general ICU-population. The study will focus on diagnostics of the different types of cardiomyopathy and differentiating between ischemic and non-ischemic left ventricular dysfunction in a general ICU population. The aim of this study is to assess the incidence and prognosis of the different types of left ventricular dysfunction in critically ill patients. Our hypothesis is that left ventricular dysfunction is common in the critically ill and is associated with an increased risk of short-term death.

ELIGIBILITY:
Inclusion Criteria:

* Admitted within 24 hours to the ICU
* Dysfunction of at least one organ system, defined as at least +1 point in SOFA-score.

Exclusion Criteria

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General ICU population
Sampling Method: Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  All cause mortality after admission to the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Jonatan Oras, MD, PhD, Principal Investigator — Sahlgrenska Academy, University of Gothenburg
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götalandsregionen, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Not decided

REFERENCES:
- [Derived] Cavefors O, Ljung Faxen U, Bech-Hanssen O, Lundin S, Ricksten SE, Redfors B, Oras J. Isolated diastolic dysfunction is associated with increased mortality in critically ill patients. J Crit Care. 2023 Aug;76:154290. doi: 10.1016/j.jcrc.2023.154290. Epub 2023 Mar 20. PMID 36947970